CLINICAL TRIAL: NCT06484439
Title: "A Prospective Randomized Controlled Trial to Determine Most Effective Post-Operative Analgesia After Third Molar Extraction"
Brief Title: Controlled Trial to Determine Most Effective Post-Operative Analgesia After Third Molar Extraction
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Principal Investigator, Patrick Morrell, Principal Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMCSD.2018.0014
Record Dates: First submitted 2024-06-04; First posted 2024-07-03 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Pain, Post-operative; Third Molar; Oral Surgery; Pain, Acute
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Ketorolac; Ketorolac Tromethamine; Oxycodone; Acetaminophen; Ibuprofen; Hydrocodone; acetaminophen, hydrocodone drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be randomly assigned to one of two groups. Each group will be given one of two post-operative medication regimens consisting of a combination of either (1) Acetaminophen (Tylenol), Oxycodone, and Ibuprofen (Motrin), or (2) Acetaminophen (Tylenol), Oxycodone, and Ketorolac (Toradol).
  This research study is a double blind study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetaminophen, Ibuprofen, Hydrocodone Control arm (Active Comparator): The control arm will be 650 mg Acetaminophen PO scheduled q6h, 600mg Ibuprofen PO scheduled q6h and 5 mg Hydrocodone PO PRN q6h.
  Interventions: Drug: Acetaminophen; Drug: Ibuprofen; Drug: Hydrocodone
- Ketorolac, Acetaminophen, Oxycodone Study arm (Experimental): The study arm will be 10 mg Ketorolac PO q6h, 650 mg Acetaminophen PO scheduled q6h, and 5 mg Oxycodone PO PRN q6h.
  Interventions: Drug: Ketorolac; Drug: Oxycodone; Drug: Acetaminophen

INTERVENTIONS:
Drug: Ketorolac — 10 mg PO q 6h scheduled
  Other Names: Toradol
  Arms: Ketorolac, Acetaminophen, Oxycodone Study arm
Drug: Oxycodone — 5 mg PO PRN
  Other Names: Oxycontin
  Arms: Ketorolac, Acetaminophen, Oxycodone Study arm
Drug: Acetaminophen — 650 mg q 6h scheduled
  Other Names: Tylenol
Drug: Ibuprofen — 600 mg PO scheduled q6h
  Other Names: Motrin
  Arms: Acetaminophen, Ibuprofen, Hydrocodone Control arm
Drug: Hydrocodone — 5 mg hydrocodone PO PRN q6h
  Other Names: Vicodin
  Arms: Acetaminophen, Ibuprofen, Hydrocodone Control arm

SUMMARY:
This is a prospective randomized clinical trial that will investigate which post-operative medications in conjunction with a multimodal analgesia approach can most effectively control post-operative pain and reduce opioid consumption.

DETAILED DESCRIPTION:
The recruitment of patients is covered in another section. Once patients are recruited based on inclusion/exclusion criteria, they will be consented and randomized into one of the 2 arms. The pre and perioperative anesthesia protocols will be identical for each arm and will consist of an opioid free general anesthesia. Local anesthesia will be given in an identical fashion in all arms. One cartridge of 2% lidocaine with 1:100k epinephrine will be given as a nerve block for the inferior alveolar nerve bilaterally. Then one cartridge of 0.5% bupivacaine with 1:200k epinephrine will be locally injected for at each of the four 3rd molar sites. Both arms will be injected with 133mg (10cc) of liposomal bupivacaine. The third molars will then be extracted in typical fashion. Each patient will be attached to one of two postoperative arms distinguished by the post-operative medications received. The control arm will be 650 mg Tylenol PO scheduled q6h, 600mg Motrin per os (PO) scheduled q6h and 5 mg hydrocodone PO pro re nata (PRN) q6h. The study arm will be 10 mg Toradol PO q6h, 650 mg acetaminophen PO scheduled q6h, and 5 mg oxycodone PO PRN q6h. The blinded medication will be either the 600mg Motrin or the 10mg Toradol. The patients will be standard 3rd molar extraction post-operative instructions as well as specific instructions on how to take medications. The identity of the patients will be linked to a key that will be kept in a locked box inside a keypad entry office. All future pain assessors will be blinded to the arm of the study in which the patient is attached. The patients will respond to daily pain intensity scores, medications taken, quality of life measures through a survey. The patients will be taught about the surveys during the consent process and again postoperatively. An email or phone will be done for the patients on the following morning for the first 5 days postoperatively. The patient will be instructed to complete the survey that will assess pain, medications taken and quality of life items. The patients will submit these daily until they return to clinic 5 days post-op where they will again submit one survey collectively discussing the outcomes of the previous 5 days. All arms will have the primary investigator's cell phone number if any adverse reactions present themselves.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 years or older
* Scheduled for 3rd molar extraction (x4) with at least one mandibular 3rd molar impacted
* American Society of Anesthesiologists classification 1 or 2
* Able to provide consent, adhere to study schedule, complete study journal, and understand English

Exclusion Criteria:

* History of hypersensitivity or idiosyncratic reaction to amide-type local anesthetics or opioids
* Contraindication to lidocaine, epinephrine, bupivacaine, or hydrocodone
* Significant drug allergy history
* Currently pregnant or nursing at time of study or within 1 month of drug administration
* Severe renal or hepatic impairment, significant cardiovascular disease; migraines, frequent headaches.
* Use of any of the following medication within 1 month of EXPAREL infiltration or if the medications are being given to control pain: Selective Serotonin Reuptake Inhibitors (SSRIs), Serotonin Nonadrenaline Reuptake Inhibitors (SNRIs), gabapentin, pregabalin, or duloxetine.
* Current use of systemic glucocorticosteroids within 1 month of enrollment in the study
* No concurrent surgical procedures within 2 weeks before or after 3rd molar extractions

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Post operative pain control after third molar extraction | Up to five days post operative procedure.
  All participants will complete a daily survey on the medications taken to relieve pain.
Post operative opioid use after third molar extraction | Up to five days post operative procedure.
  Daily survey will be used to assess the amount of post operative opioid us including dosage and frequency of use.
Post operative pain assessment after third molar extraction | Up to five days post operative procedure.
  Participants fill out daily for five days post operative procedure the Numeric Pain Rating Scale (NPRS). This is a ten point scale with 0 = No pain, 5 = Moderate pain, 10 = Worst possible pain. The higher the number is a worse outcome.
Post operative quality of life assessment after third molar extraction | Up to five days after third molar extraction.
  Post operative quality of life was ascertained with the 10 point Likert scaled question, "What is your rating for your actual overall comfort?'. 1 = Very low overall comfort, 5 = Neither low or high overall comfort, 10 = Very high overall comfort.
  The higher the score means a better outcome. This question is part of the daily survey that participants filled out for five days post operative procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick T Morrell, DMD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Naval Medical Center San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No